CLINICAL TRIAL: NCT02777645
Title: Growth, Dietary Intakes and Feeding Behaviors of Children With Cerebral Palsy Who Have Chewing Disorders
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, PT, PhD, Hacettepe University
Other Study IDs: ArslanSerel1
Record Dates: First submitted 2016-05-13; First posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Cerebral Palsy; Mastication Disorder; Malnutrition; Growth Delay
MeSH Terms: conditions — Cerebral Palsy; Malnutrition | interventions — Growth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group: Study group(n=50) included CP children with chewing disorder. Growth, feeding evaluation will be done.
  Interventions: Other: Growth, feeding evaluation
- Control group: Control group(n=35)= healthy children without chewing disorder Growth, feeding evaluation will be done.
  Interventions: Other: Growth, feeding evaluation

INTERVENTIONS:
Other: Growth, feeding evaluation — Z-scores of the nutritional indicators were calculated. The dietary assessment was performed by using the 24-hour recall method. The Behavioural Paediatrics Feeding Assessment Scale (BPFAS) was used to assess both frequencies of negative feeding behaviours and parents' problematic perceptions

SUMMARY:
The nutritional status of CP children may be decreased when children have chewing disorders too due to insufficient solid food intake. The objective of this study was to investigate growth, dietary intakes and feeding behaviours of children with CP who have chewing disorders, and to compare them with their healthy peers.

DETAILED DESCRIPTION:
Chewing function is defined as a rhythmic oral motor activity to comminute and soften solid food. Children with CP often have difficulty in transitioning to solid food. The main food of 45% of them was liquids and semisolids. It was reported that food/fluid textures were modified for 39% of children in which with poorer gross motor function tended to receive a greater proportion of energy from fluids in their diets and fewer chewable foods. Lopes et al. investigated dietary patterns of 90 children with CP aged 2-13 years by using the 24-hour recall method and found that 26% and 9% of children had difficulty in chewing and swallowing of solid foods, respectively. However, the diet of children with normal feeding skills includes liquid, semisolid and/or solid foods together so unable to take any solid food may affect sufficient food intake and nutritional status of children with CP who have chewing disorders. The significance of this situation is that nutritional status has effects on general health and quality of life of children and their families. Therefore, it is important to show the nutritional status of CP children with chewing disorders to increase the awareness of both parents and healthcare providers on solid food intake and solve the problem early. The objective of this study was to investigate growth, dietary intakes and feeding behaviours of children with CP who have chewing disorders, and to compare them with their healthy peers.

ELIGIBILITY:
Inclusion Criteria:

Study group

* Children with cerebral palsy
* Having complaints about chewing function
* Do not manage solid food intake
* Above the age of 18 months Control group
* Healthy children
* No complaints about chewing function
* Can manage solid food intake
* Above the age of 18 months

Exclusion Criteria:

* Under the age of 18 months
* Requiring tube feeding or taking any oral nutritional supplements
* Using any medicine and/or oral appliances that could affect the chewing performance

Ages: 24 Months to 61 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Group I (study group) (n=50) included CP children with chewing disorders and group II (control group) (n=35) included healthy children without chewing disorders
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Growth of children with cerebral palsy (CP) who have chewing disorders (Z-scores) | 3 months
  Z-scores of the nutritional indicators were calculated.

SECONDARY OUTCOMES:
Dietary intakes of children with cerebral palsy (CP) who have chewing disorders (dietary assessment) | 3 months
  The dietary assessment was performed by using the 24-hour recall method.
Feeding behaviours of children with cerebral palsy (CP) who have chewing disorders (BPFAS) | 3 months
  The Behavioural Paediatrics Feeding Assessment Scale (BPFAS) was used to assess both frequencies of negative feeding behaviours and parents' problematic perceptions.

CONTACTS AND LOCATIONS:
Overall Officials: Selen SEREL ARSLAN, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacetttepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided